CLINICAL TRIAL: NCT06463652
Title: Cervical Cerclage With Vaginal Progesterone Versus Vaginal Progesterone Only for Preterm Birth Prevention in Women With a Singleton Pregnancy and a Short Cervical Length: a Randomized Clinical Trial
Brief Title: Cerclage With Progesterone Versus Progesterone Only in Singleton Pregnancies
Acronym: RESILIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08/24/DD-BVMD
Record Dates: First submitted 2024-06-07; First posted 2024-06-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Preterm Birth; Short Cervix
Keywords: Cerclage; Progesterone; Singleton; Preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined therapy group (cervical cerclage plus vaginal progesterone) (Experimental): Women will be receiving the cervical cerclage according to local protocol within a week after randomization, using the McDonald technique.
  Within one day after the procedure, they will be receiving 200 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 200mg, Actavis, United Kingdom), once daily at bedtime. Participants will be asked to record their drug application in a patient diary sheet.
  Interventions: Procedure: Cervical cerclage; Drug: Vaginal progesterone
- Progesterone only group (Active Comparator): Women allocated to the progesterone only group will be receiving 200 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 200mg, Actavis, United Kingdom), once daily at bedtime. Participants will be asked to record their drug application in a patient diary sheet.
  Interventions: Drug: Vaginal progesterone

INTERVENTIONS:
Procedure: Cervical cerclage — Cervical cerclage using the McDonald technique under anaesthesia.
  Arms: Combined therapy group (cervical cerclage plus vaginal progesterone)
Drug: Vaginal progesterone — Cyclogest® 200mg, Actavis, United Kingdom, applied once daily at bedtime.
  Other Names: Cyclogest® 200 mg

SUMMARY:
This study compares the effectiveness of cervical cerclage with vaginal progesterone to vaginal progesterone only for the prevention of preterm birth in women with a singleton pregnancy and a short cervical length. Participants will be randomly assigned in a 1:1 ratio to receive cerclage plus progesterone or progesterone only.

DETAILED DESCRIPTION:
This open-label, multi-center, randomized controlled trial aims to compare the effectiveness of cervical cerclage with vaginal progesterone (the combined therapy group) to vaginal progesterone only (the progesterone-only group) for the prevention of preterm birth in women with a singleton pregnancy and a cervical length ≤ 25mm.

After written informed consent, women will be randomly assigned in a 1:1 ratio to receive a cervical cerclage with vaginal progesterone or vaginal progesterone only. Randomization will be carried out by entering participant details into HOPE Epi® (a web portal of HOPE Research Center, My Duc Hospital). Treatment allocation will be assigned according to a computer-generated randomization list stored in the online system, with a permuted random block size of 2, 4, or 6. Blinding will not be possible due to the nature of interventions. However, neonatologists assessing the neonates will be unaware of treatment allocation. Apart from randomization, participants will be monitored and treated according to local protocol.

All women at 16 0/7 to 24 0/7 weeks' gestation with a singleton pregnancy will undergo cervical length measurement and digital examination at screening routinely. Women with a cervical length ≤25 mm will be eligible for the study. Eligible women will further undergo a speculum examination to assess the feasibility of treatment with either cervical cerclage or vaginal progesterone and to exclude premature rupture of the membranes, acute vaginitis, and cervicitis. Only women in whom the clinician assesses both treatments as feasible will be randomized.

Women allocated to a combined therapy group will receive the intervention according to local protocol within a week after randomization. Briefly, cervical cerclage (McDonald technique) will be performed in the operation theatre. From the same day of undergoing cerclage, participants will be receiving 200 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 200mg, Actavis, United Kingdom), once daily at bedtime. Participants will be asked to record their drug application in a participant diary sheet.

Women allocated to the progesterone-only group will be receiving 200 mg vaginal progesterone, purchased from the manufacturer (Cyclogest® 200mg, Actavis, United Kingdom), once daily at bedtime. Participants will be asked to record their drug application in a participant diary sheet.

In both groups, interventions will be stopped at 37 0/7 weeks of gestation or at delivery.

Primary analysis will be performed on an intention-to-treat basis. The primary outcome, the time from randomization to delivery, will be summarised as median and IQR and compared between the two arms using the Mann-Whitney test. A mean ratio with a 95% confidence interval will be calculated to assess the effect of the treatment. Kaplan-Meier and Cox proportional hazard analysis will be performed in which the gestational week at delivery will be the time scale, continued pregnancy will be the event, and results will be compared with a log-rank test. Hazard ratio (HR) values will be estimated using a Cox proportional hazards model, with a formal test of the proportional hazard assumption.

The secondary outcome will be analysed by reporting continuous variables as mean and standard deviation for normally distributed variables or median and interquartile range (Q1; Q3) for non-normally distributed variables. Categorical variables will be presented as the number of events and proportions. Student T-test or Mann-Whitney U test will be used for continuous outcomes to compare the differences between groups. For categorical outcomes, the Chi-squared or Fisher exact test will be used. In the case of dichotomous endpoints, the relative risk (RR) and 95% confidence interval (CI) values will be calculated using the Wald or Adjusted Wald methods for a small proportion. Per-protocol analysis will also be conducted if needed.

A prespecified subgroup analysis will be performed by quartiles of cervical length, which tested for interaction between cervical length and the treatment effect on the primary outcome, the major secondary outcome and PTB <28, <34, <37 weeks.

The p-values <0.05 will be considered to indicate statistical significance. Statistical analyses will be performed using the R statistical software.

Details of the analysis will be described in a separate statistical analysis plan developed during the study and finalized before the data lock. Cost data will be collected and will be reported on a separated paper.

Interim analysis will be done after completion of data recruitment of the first 162 participants, by an independent Data Safety Monitoring Committee. The Data Safety Monitoring Committee will be asked to assess the primary endpoint for effectiveness. Also, the Data Safety Monitoring Committee will be provided insight into the serious adverse events (SAEs) that have occurred. The interim analysis will be conducted using a two-sided significant test with the Haybittle-Peto spending function and a type I error rate of 5 percent with p <0.001 (Z alpha = 3.29) being a reason to stop the trial. The continuation of the study will depend on the advice of Data Safety Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥18 years
* Singleton pregnancy
* Cervical length ≤ 25 mm, measured by TVS at the second-trimester ultrasonography (16 0/7 - 24 0/7 weeks of gestation)
* Not participating in any other study which has intervention on maternity or fetus
* Provision of written informed consent as shown by a signature on the participant consent form.

Exclusion Criteria:

* Cervical dilation with visible amniotic membranes or amniotic membranes prolapsed into the vagina
* Major congenital abnormalities of the fetus
* Intrauterine fetal demise
* Presence of severe vaginal discharge*
* Presence of vaginitis or cervicitis*
* Presence of vaginal bleeding*
* Placenta previa or vasa previa
* Preterm premature rupture of membranes
* Preterm labor without ruptured membrane at the time of screening
* Suspected chorioamnionitis
* Unable to undergo cerclage
* Cerclage in place
* Allergy to progesterone

(*Women with acute cervicitis, vaginitis or severe vaginal discharge are eligible once they have been treated and if they have a CL ≤25 mm between 16 0/7 - 24 0/7 weeks of gestation.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to delivery | From date of randomization until the date of delivery
  Number of days between randomization and delivery

SECONDARY OUTCOMES:
Composite poor neonatal outcomes (major sencondary endpoint) | From 20 weeks of gestation to 28 days after estimated due date
  Stillbirth or neonatal death, intraventricular haemorrhage, respiratory distress syndrome, necrotizing enterocolitis or neonatal sepsis.
Miscarriage <22 weeks (late miscarriage) | From date of randomization to 22 weeks of gestation
  spontaneous loss of pregnancy between 12 to 22 weeks is termed as late miscarriage
Gestational age at delivery | At delivery
  Gestational age at delivery
Preterm birth <24 weeks, <28 weeks, <32 weeks, <34 weeks and <37 weeks of gestation | At delivery
  Preterm birth is defined as any birth ≥ 22 and < 37 completed weeks of gestation. Any birth < 22 weeks is defined as late miscarriage
Spontaneous preterm birth <24 weeks, <28 weeks, <32 weeks, <34 weeks and <37 weeks of gestation | At delivery
  Spontaneous preterm birth, including preterm labour, preterm spontaneous rupture of membranes, preterm premature rupture of membranes, and cervical weakness before 24 weeks, 28 weeks, 32 weeks, 34 weeks, and 37 weeks of gestation, respectively, does not include indicated preterm delivery for maternal or fetal conditions.
Iatrogenic preterm birth <24 weeks, <28 weeks, <32 weeks, <34 weeks and <37 weeks of gestation | At delivery
  Iatrogenic preterm birth, including planned delivery that occurs before 24 weeks, 28 weeks, 32 weeks, 34 weeks, and 37 weeks of gestation, respectively, due to maternal and/or fetal causes.
Onset of labor | At birth
  Classified as spontaneous, labor induction, or elective C-section.
Mode of delivery | At birth
  Classified as vaginal delivery or C-section (elective, suspected fetal distress, non-progressive labor).
Live birth | At birth
  Defined as the complete expulsion or extraction from a woman of a product of fertilization after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown
Use of tocolytic drugs | From 24 0/7 to 33 6/7 weeks' gestation
  Use of any tocolytic drug to treat preterm labour
Use of Post cerclage antibiotics | Within one week after the cerclage procedure
  Use of any treatment antibiotics after the cerclage procedure
Use of antenatal corticosteroids | From 24 0/7 to 33 6/7 weeks' gestation
  Use of antenatal corticosteroids to prevent respiratory distressed syndrome
Use of MgSO4 for neuroprotection | From 24 0/7 to 31 6/7 weeks' gestation
  Use of MgSO4 for neuroprotection
Fetal growth restriction | From randomization to delivery
  It is defined as the failure of the fetus to meet its growth potential due to a pathological factor, most commonly placental dysfunction.
Preterm premature rupture of membranes | From randomization to before 37 weeks of gestation
  When membrane rupture occurs before labor and before 37 weeks of gestation
Length of maternal admission for labour | Up to 2 weeks after birth
  Number of maternal admission days for labour
Total length of admission for threatened preterm labor | From 22 0/7 to 36 6/7 weeks of gestation
  Number of admission days for treatment of preterm labour
Chorioamnionitis | From randomization to delivery
  Intraamniotic infection (diagnosed according to The American College of Obstetricians and Gynecologists Committee on Obstetric Practice No 712, 2017 (reaffirmed 2022))
Maternal mortality | From randomization to during pregnancy and childbirth or within 42 days of termination of pregnancy
  female deaths from any cause related to or aggravated by pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy
Maternal side effects | From date of randomization until delivery
  Vaginal discharge, vaginal bleeding, vaginal infection (confirmed by vaginal discharge culture), preterm premature rupture of membranes, chorioamnionitis, necrosis or rupture of the cervix, cervical laceration, vaginal or bladder injury.
Birthweight | At birth
  Weight of the newborn measured right after delivery
Birthweight <1500 g | At birth
  Weight of the newborn <1500g
Birthweight <2500 g | At birth
  Weight of the newborn <2500g
Congenital anomalies | After randomization to at birth
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally and at birth. Congenital anomalies can be caused by single gene defects, chromosomal disorders, multifactorial inheritance, environmental teratogens, and micronutrient deficiencies. The time of identification will be reported.
1-min Apgar score | 1 min after birth
  Apgar score at 1 minute after birth
5-min Apgar score | 5 min after birth
  Apgar score at 5 minute after birth
Admission to neonatal intensive care unit | At birth and up to 28 days after birth
  Admission to neonatal intensive care unit of baby
Length of stay in the neonatal intensive care unit | Up to 28 days after estimated due date
  Number of admission days to neonatal intensive care unit
Neonatal death | Within the first 28 days of life after delivery
  Death of a live-born baby within 28 days of birth
All stillbirth | After 20 weeks of gestation
  Defined as the death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles. It includes deaths occurring during labor.
  All stillbirth will be defined as a baby born with no signs of life at ≥ 20 weeks of gestation
Early stillbirth | ≥ 20 weeks and < 28 weeks of gestation
  A baby born with no signs of life at ≥ 20 weeks and < 28 weeks of gestation
Late stillbirth | After 28 weeks of gestation
  A baby born with no signs of life at ≥ 28 weeks of gestation
Perinatal death | From 20 weeks of gestation to the first 28 days of life after delivery
  Either stillbirth or neonatal death
Respiratory distress syndrome | Up to 28 days after estimated due date
  Diagnosed as the presence of tachypnoea >60/minute, sternal recession and expiratory grunting, need for supplemental oxygen, and a radiological picture of diffuse reticulogranular shadowing with an air bronchogram
Intraventricular haemorrhage II B or worse | Up to 28 days after estimated due date
  Diagnosed by repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al
Necrotizing enterocolitis | Up to 28 days after estimated due date
  An acquired gastrointestinal disease associated with significant morbidity and mortality in prematurely born neonates. Necrotizing enterocolitis will be diagnosed according to Bell et al., 1978
Neonatal sepsis | Up to 28 days after estimated due date
  Diagnosed on the combination of clinical signs and positive blood cultures of the newborn

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No